CLINICAL TRIAL: NCT01328080
Title: Improving Acne Keloidalis Nuchae by Inducing Matrix Metalloproteinases in Vivo Using Targeted Ultraviolet-B Irradiation
Brief Title: Treatment of Acne Keloidalis Nuchae (Razor Bumps Behind the Neck) Using UV Light Therapy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: Skin of Color Society (Unknown)
Responsible Party: Principal Investigator, Ginette Okoye, MD, Assistant Professor, Johns Hopkins University
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: NA_00035842
Record Dates: First submitted 2011-03-31; First posted 2011-04-04 (Estimated); Results first posted 2014-06-16 (Estimated); Last update posted 2017-03-29 (Actual); Status verified 2017-02

CONDITIONS: Acne Keloidalis Nuchae
MeSH Terms: conditions — Acne Keloid

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Targeted UV-B (Left) (Experimental): Targeted UV-B on left side of the scalp.
  Interventions: Radiation: Targeted UV-B
- Targeted UV-B (Right) (Experimental): Targeted UV-B on right side of the scalp.
  Interventions: Radiation: Targeted UV-B

INTERVENTIONS:
Radiation: Targeted UV-B — Daavlin Lumera phototherapy device (290-320 nm), dosed by patients' individual minimal erythema dose (MED)

SUMMARY:
This study is being done to evaluate the effect of targeted UV-B (a component of sunlight) on the treatment of acne keloidalis nuchae (AKN, or razor bumps on the back of the neck). The investigators believe targeted UV-B is a safe and effective way to reduce the appearance of AKN.

ELIGIBILITY:
Inclusion Criteria:

* age 18 or over
* male gender
* African-American or other black ethnicity
* current diagnosis of acne keloidalis nuchae (razor bumps on back of neck)

Exclusion Criteria:

* allergy to lidocaine or numbing medicine
* history of increased sensitivity to sunlight, lupus, or porphyria
* current use of a drug that increases sensitivity to sunlight

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2011-02; Primary Completion 2012-08 (Actual); Study Completion 2012-08 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Johns Hopkins Dept. of Dermatology, Baltimore, Maryland, United States

REFERENCES:
- See also: Skin of Color Society (sponsor) — http://www.skinofcolorsociety.org/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from patient populations evaluated by the Johns Hopkins Department of Dermatology located at the Johns Hopkins Outpatient Center between April 2011 through April 2012. Participants were also be recruited from other patient populations at the Johns Hopkins Hospital through the use of advertisements.
Pre-assignment Details: Prior to UVB treatment,each subject's Minimal Erythema dose (MED) was determined. Exclusion criteria: photosensitive disorders,skin cancer,previous radiation therapy,use of photosensitizing drugs,lidocaine allergy,bleeding disorders,pregnancy,and lactation. Wash out: 4 weeks for antibiotics/corticosteroids, 6 months for oral isotretinoin.
Groups:
- Targeted UVB Phototherapy: All patients were randomly assigned to receive targeted UVB phototherapy 3 times a week for 16 weeks to either the right or the left side of the scalp. The untreated side served as an internal control until the end of week 8, after which both sides of the scalp were treated.
Period: Overall Study
Arm/Group | Targeted UVB Phototherapy
Started | 11 (11 subjects consented; 1 withdrew consent before first UVB treatment)
Completed | 6
Not Completed | 5
Not completed — Lost to Follow-up | 5

BASELINE CHARACTERISTICS:
Arm/Group | Targeted UV-B
Number analyzed (Participants) | 11
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 11
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 36.6 (6.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 11
Region of Enrollment [Number; unit: participants]
  United States | 11

OUTCOME MEASURES:

1. Primary Outcome: Percentage Change in Total AKN Lesions From Baseline to Week 16.
Description: To determine if treatment of AKN with targeted ultraviolet B radiation will improve the clinical appearance of lesions.
Time Frame: Baseline to Week 16
Measure: Mean (Full Range); unit: percentage of lesion count reduction
Arm/Group | Targeted UVB Phototherapy
Number analyzed (Participants) | 6
percentage of lesion count reduction | 49 [29 to 61]

ADVERSE EVENTS:
Time Frame: 16 weeks
Arm/Group | Targeted UVB Phototherapy
Serious Adverse Events (participants affected / at risk) | 0/11
Other Adverse Events (participants affected / at risk) | 2/11
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Targeted UVB Phototherapy (N=11)
erythema (Skin and subcutaneous tissue disorders) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No